CLINICAL TRIAL: NCT02230449
Title: Identifying Markers of Oocyte Competence Through a Maturation Analysis
Brief Title: Identifying Expression Markers of Cumulus Cells to Identify Oocyte Developmental Potential Through a Maturation Analysis
Status: Completed | Type: Observational
Sponsor: Memorial Sisli Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Prof. Dr. Semra Kahraman, Director of ART and Genetics Center, Memorial Sisli Hospital, Istanbul
Other Study IDs: OocyteCompetenceSK001; GFI-2014-#21 (Other Grant/Funding Number: Merck Serono Grant For Fertility Innovation)
Record Dates: First submitted 2014-08-19; First posted 2014-09-03 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cumulus cells from each oocyte of every enrolled patient will be collected and mRNA & miRNA extraction will be performed.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to analyze the expression of genes and microRNAs potentially involved in oocyte competence in follicles of different sizes (<17mm and ≥17mm) at the time of oocyte pick-up.

DETAILED DESCRIPTION:
In ART, one of the major obstacles encountered in some patients is the wide variation in the follicular size at the oocyte pick-up day and consequently, the number of available mature oocytes and the number of competent embryos for implantation. The follicular size at the day of oocyte pick-up reflects the synchronicity of the individual follicular responsiveness to FSH.

For successful preimplantation development of an embryo, the oocyte must contain all necessary maternal factors. Two of these factors are specific mRNA transcripts (GDF9, PTX3, HAS2, PTGS2, TNFAIP6) and microRNA (miR-224).

For each Cumulus Oocyte Complex, the evaluation of embryo development and morphokinetics will be correlated with the expression and implantation data to identify a quantitative biomarker to predict the embryo with the highest chance of implantation in patients.

Experimental Design:

1. - Collection of Cumulus Oocyte Complex (COC) from patients
2. - Separation of oocytes according to the size of the follicule they have been retrieved from (<17mm; ≥17mm)
3. - Isolation of mRNA from both groups of cumulus cells
4. - Expression studies, qRT-PCR (GDF9, PTX3, HAS2, PTGS2, TNFAIP6)
5. - Analysis of miR-224, a negative regulator of cumulus expansion via PTX3
6. - Time-lapse culture & evaluation of morphokinetics

ELIGIBILITY:
Inclusion Criteria:

* No more than 2 previous treatment cycles
* No history of recurrent spontaneous abortions
* Age ≤ 39 years
* BMI < 30 kg / m2
* ≥ 8 cumulus-oocyte-complexes (COC) retrieved
* human Chorionic Gonadotrophin (hCG) triggering

Exclusion Criteria:

* Preimplantaion Genetic Diagnosis (PGD) or Preimplantation Genetics Screening (PGS) indication
* Maximum number of 24 COC during pickup
* Failure to culture until Day 5
* Polycystic ovary syndrome
* Severe endometrial factor that can influence implantation
* Uterine malformation or congenital anomaly
* Severe male factor (Azoospermia)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile couples applying to the clinic for assisted reproductive technologies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cumulus cell RNA expression correlation with blastocyst formation potential and quality | 6 days
  At the day of oocyte pick-up, cumulus cells will be collected from each cumulus oocyte complex. RNA extraction will be performed from those cumulus cells and expression levels of 5 genes and 1 miRNA will be measured (compared with that of a housekeeping gene). Oocytes of those samples will be injected and cultured with routine Assisted Reproduction Techniques. At the day 5 & 6, after the oocyte pick-up procedure, each blastocyst formed will be noted and the quality of each blastocyst will be recorded. The blastocyst grading will be done according to Gardner's blastocyst morphological criteria (degree of expansion of the blastocoele cavity: 1 to 5, inner cell mass morphology: A to C, trophectoderm morphology: A to C).
  The composite primary outcome measure will allow the correlation of the expression levels of 5 genes and 1 miRNA of each cumulus oocyte complex with the corresponding embryo morphology on day 5 (presence or absence of a blastocyst) and blastocyst quality.

SECONDARY OUTCOMES:
Implantation Rate | 2 months
  Implantation of the embryo(s) transferred will be checked by ultrasound 6 weeks after the pick-up. Patients for whom the number of embryo(s) transferred match the number of sac will allow the correlation of the expression data with implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Kahraman, Prof. Dr, Study Chair — Manager of ART and Genetics Center; Semra Kahraman, Prof. Dr., Study Director — Manager of ART and Genetics Center; Mehmet Ali Tufekci, PhD, Principal Investigator — ART Center Research and Development Department
Locations (1):
- Memorial Sisli Hospital ART Center, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Kahraman S, Cetinkaya CP, Cetinkaya M, Tufekci MA, Ekmekci CG, Montag M. Is there a correlation between follicle size and gene expression in cumulus cells and is gene expression an indicator of embryo development? Reprod Biol Endocrinol. 2018 Jul 21;16(1):69. doi: 10.1186/s12958-018-0388-0. PMID 30031399